CLINICAL TRIAL: NCT06639048
Title: Is There a Relationship Between Individuals' Social Media Use and Their Fears of Eating Disorders?
Brief Title: Social Media and Eating Disorder Fear
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Rahime Evra KARAKAYA, Principal Investigator, Ankara Yildirim Beyazıt University
Other Study IDs: AnkaraYBU-KARAKAYA003
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Eating Disorder; University Students; Social Media; Eating Behavior; Fear
Keywords: social media; eating disorder; fear
MeSH Terms: conditions — Feeding and Eating Disorders; Feeding Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University students: Those with using social media
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire including demographic characteristics, social media usage habits, body weight, height, effects of social media on eating behavior scale and eating disorder fear questionnaire.

SUMMARY:
The goal of this observational study is to learn about the relationship between social media use and fear of eating disorders in university students. The main question it aims to answer is:

Is there a relationship between social media use and eating disorder fears in university students?

University students will answer a questionnaire face to face, including questions about their social media usage habits, the impact of social media on eating behavior scale, and the fears of eating disorders scale.

ELIGIBILITY:
Inclusion Criteria:

* Using social media

Exclusion Criteria:

* Pregnant or lactating individuals

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ankara Yıldırım Beyazıt University, Faculty of Health Sciences students
Sampling Method: Non-Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Social media usage habits | Baseline
  number and percentage
Eating Disorder Fear Questionnaire | Baseline
  The Eating Disorder Fear Questionnaire is a tool designed to measure individuals' fears related to eating disorders. The Turkish validity and reliability of the scale were conducted by Kahraman and Kerimler in 2021. The scale is in a 7-point Likert format, with a minimum score of 17 and a maximum score of 119. Higher scores on both the sub-dimensions and the overall scale indicate greater fears related to eating disorders.
Effects of social media on eating behavior scale | Baseline
  The scale developed by Alev Keser consists of 18 items in a unidimensional 5-point Likert format (Never-1 point, Rarely-2 points, Sometimes-3 points, Often-4 points, Always-5 points). The scores obtained from the responses are summed, with a minimum score of 18 and a maximum score of 90. As the score increases, it indicates a greater influence of social media on eating behavior.

SECONDARY OUTCOMES:
Demographic characteristics | Baseline
  number and percentage
Body weight | Baseline
  Body weight in kg
Height | Baseline
  Height in cm

CONTACTS AND LOCATIONS:
Overall Officials: Rahime E Karakaya, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No